CLINICAL TRIAL: NCT00184119
Title: Effects of a Psychiatric Intensive Care Unit in an Acute Psychiatric Department.
Brief Title: Effects of a Psychiatric Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AEV-01
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Mental Disorders
Keywords: Emergency services, psychiatric; Intensive care units; Hospitals, psychiatric; Aggression; Violence
MeSH Terms: conditions — Mental Disorders; Aggression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychiatric Intensive Care Unit (Experimental)
  Interventions: Procedure: Psychiatric Intensive Care Unit
- Whole acute unit (Active Comparator)
  Interventions: Procedure: Care in whole acute unit

INTERVENTIONS:
Procedure: Psychiatric Intensive Care Unit
  Arms: Psychiatric Intensive Care Unit
Procedure: Care in whole acute unit — psychiatric acute care as usual
  Arms: Whole acute unit

SUMMARY:
The purpose of the study is to compare the effects of using or not using a Psychiatric Intensive Care Unit (PICU) in an acute psychiatric department.

DETAILED DESCRIPTION:
The main aim of the study is to compare the effects of using or not using a Psychiatric Intensive Care Unit (PICU) in an acute psychiatric department.The acute ward of Østmarka psychiatric department, St. Olavs Hospital has a PICU separated from the rest of the ward. The PICU is separated with a locked door. Under two different conditions at different times all patients evaluated to be in need of PICU were admitted to the PICU. In the first condition the doors inside the PICU and between the rest of the acute ward and PICU were closed or locked. In the second condition the doors inside the PICU and the door between the PICU and the rest of the acute ward were either removed or held permanently open. In the second condition the patients thus were admitted to a PICU unit not using PICU principles.

The patients were evaluated with different rating scales at admittance, day three and at discharge from PICU.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to Østmarka psychiatric department, St. Olavs Hospital in need of a PICU.

Exclusion Criteria:

* Patients with dementia or mental retardation to an extensive degree.
* Patients not speaking Norwegian or English.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2001-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Length of stay in Psychiatric Intensive Care Unit (PICU) | 3 days
Symptoms of psychopathology | 3 days
  assessed by Broset Violence Checklist (BVC), a six-item observer-rated scale scoring behaviours. Higher scores predict imminent violence in psychiatric inpatients
Violent or threatening incidents | 3 days
  recorded with the Staff Observation Aggression Scale-Revised (SOAS-R),

SECONDARY OUTCOMES:
Therapeutic steps and nurses' interventions | 3 days
  coded daily on a 23-item checklist

CONTACTS AND LOCATIONS:
Overall Officials: Olav M Linaker, Professor, Study Chair — Norwegian University of Science and Technology
Locations (1):
- Østmarka Psychiatric Department, St. Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vaaler AE, Morken G, Flovig JC, Iversen VC, Linaker OM. Effects of a psychiatric intensive care unit in an acute psychiatric department. Nord J Psychiatry. 2006;60(2):144-9. doi: 10.1080/08039480600583472. PMID 16635934
- [Derived] Vaaler AE, Iversen VC, Morken G, Flovig JC, Palmstierna T, Linaker OM. Short-term prediction of threatening and violent behaviour in an Acute Psychiatric Intensive Care Unit based on patient and environment characteristics. BMC Psychiatry. 2011 Mar 18;11:44. doi: 10.1186/1471-244X-11-44. PMID 21418581